CLINICAL TRIAL: NCT01366781
Title: Effects of Varying Meal Size on Gut Hormone and Islet Hormone Secretion in Males Versus Females
Brief Title: Gut Hormones After Meal Ingestion in Males Versus Females
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lund University (Other)
Responsible Party: Principal Investigator, Bo Ahren, Professor, Lund University
Allocation: Non-Randomized | Model: Factorial | Masking: None
Other Study IDs: 004
Record Dates: First submitted 2011-05-31; First posted 2011-06-06 (Estimated); Last update posted 2014-09-30 (Estimated); Status verified 2014-09

CONDITIONS: Normal Non-fluency
Keywords: Gut hormones; Insulin secretion

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Healthy males (Experimental): Meal ingestion in healthy males
  Interventions: Other: Meal ingestion
- Healthy females (Experimental): Meal ingestion in healthy females
  Interventions: Other: Meal ingestion

INTERVENTIONS:
Other: Meal ingestion — Meal 511 kcal, meal 743 kcal or meal 1034 kcal

SUMMARY:
The study hypothesis is that the release of gut hormones is increased proportionally to caloric load in each meal. Three different meals with different meal size will therefore be served and gut hormones determined.

DETAILED DESCRIPTION:
In healthy males and females, meals with 511, 743 and 1034 kcal will be given orally. Samples will be taken during the following 300 min and gut hormones (glucose-dependent insulinotropic polypeptide and glucagon-like peptide-1) will be determined along with insulin and glucagon levels.

ELIGIBILITY:
Inclusion Criteria:

* Healthy status

Exclusion Criteria:

* Diabetes
* Liver disease
* kidney disease
* thyroid disease

Ages: 20 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2011-05; Primary Completion 2014-02 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Release of gut hormones | 300 min

SECONDARY OUTCOMES:
Insulin secretion | 300 min

CONTACTS AND LOCATIONS:
Overall Officials: Bo Ahrén, PhD, Principal Investigator — Lund University
Locations (1):
- Department of Clinical Sciences Lund, Lund University, Lund, Sweden

REFERENCES:
- [Derived] Alsalim W, Omar B, Pacini G, Bizzotto R, Mari A, Ahren B. Incretin and islet hormone responses to meals of increasing size in healthy subjects. J Clin Endocrinol Metab. 2015 Feb;100(2):561-8. doi: 10.1210/jc.2014-2865. Epub 2014 Nov 6. PMID 25375983